CLINICAL TRIAL: NCT03714659
Title: Clinical Evaluation of Autologous Micro-fragmented Adipose Tissue as a Treatment Option for Meniscus Tears
Brief Title: Autologous, Micro-fragmented Adipose Tissue for Meniscal Tears
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Jersey Regenerative Institute, LLC (Industry)
Responsible Party: Principal Investigator, Gerard Malanga, Principal Investigator, New Jersey Regenerative Institute, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-MN-201
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Tibial Meniscus Injuries; Osteoarthritis, Knee
MeSH Terms: conditions — Tibial Meniscus Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Group will receive a single injection of autologous, micro-fragmented adipose tissue into the torn meniscus and knee joint. The group will then be followed for one year, filling out pain and function questionnaires.
  Interventions: Device: Lipogems

INTERVENTIONS:
Device: Lipogems — Lipogems is a closed-loop system designed to break up adipose tissue into micro-fragmented adipose tissue without additives; therefore, meeting FDA requirements for minimal manipulation. A small volume of adipose tissue is harvested from the abdomen, thigh, or other location. The lipoaspirate is fed into the device through a reduction filter, and is then cleansed of blood and oil residues using a sterile saline solution. This fat-saline solution is then shaken for 30 seconds in a device containing stainless steel ball bearings, which further fragments and washes the lipoaspirate. Once the tissue is purified and fragmented, it is collected in 10cc sterile syringes and subsequently injected into the meniscus and knee joint.

SUMMARY:
The menisci of the knee are essential fibro-cartilaginous structures that contribute in static weight bearing, distributing compressive forces during joint movement, joint lubrication, joint stabilization, and proprioception. The menisci are commonly torn, interfering with these vital functions, with an estimated mean annual incidence as high as 60-70 per 100,000 knee injuries. When torn, the odds of developing future osteoarthritis within 2 years of follow-up can be as high as 5.92. The management of meniscal tears remains a challenge given the poor intrinsic healing capacity of tears occurring in the inner, avascular, portion of the meniscus where direct surgical repair techniques are commonly unsuccessful. Autologous adipose tissue injection has recently emerged as a promising new treatment for joint pain and soft tissue injury. Adipose can be used to provide cushioning and filling of structural defects and has been shown to have an abundance of bioactive elements and regenerative perivascular cells (pericytes).The aim of this study is to explore the potential of Lipogems® micro-fragmented adipose tissue as a meaningful treatment option for meniscus tears. Patients treated with MFAT with intra-meniscal injections under continuous ultrasound guidance are expected to report clinically meaningful improvements in knee pain and knee function after one year. Knee pain and function will be measured using a numerical pain scale (NPS) and the Knee Injury and Osteoarthritis Outcome Scale (KOOS).

DETAILED DESCRIPTION:
This is a prospective pilot study to evaluate the safety and efficacy of autologous, micro fragmented adipose tissue (Lipogems®) injection under continuous ultrasound guidance for knee pain secondary to meniscal tear(s). 20 subjects will be enrolled who present for evaluation and treatment of knee pain with associated meniscal tear despite prior conservative management. Failure of conservative management was defined as persistent pain despite the use of anti-inflammatory or other medications for pain, physical therapy, corticosteroid injections, or hyaluronic acid injections. This also included patients who were told that they were a candidate for arthroscopic surgery by an orthopedic surgeon due to failure of conservative measures. Micro-fragmented adipose tissue will be obtained by using a minimal manipulation technique in a closed system (Lipogems®), without the addition of enzymes or any additives. 1-2 mLs of micro-fragmented adipose tissue will be injected directly into visualized meniscal tears using continues ultrasound guidance. The remaining injectate will be administer into the knee joint by lateral suprapatellar approach. Post-injection guidelines including weight bearing restrictions--non-weightbearing with crutches for one week, then weight bearing as tolerated for simple daily activities--refraining from running and jumping activities and refraining from repetitive flexion beyond 90 degrees for 4 weeks total. If there was no significant pain, swelling, joint-line tenderness, and near full range of motion, unrestricted activities were allowed at the 6-8-week time-frame. Complications of both the harvest and injection sites were recorded via questionnaire at 1 and 4-week follow-up. Subjects were seen for initial follow-up at 4 weeks. They then completed surveys at 3, 6, and 12 months, including the Knee Injury and Osteoarthritis Outcome Scale (KOOS) subscales and the numerical pain scale (NPS). The NPS is one of the most common measures of pain intensity and is used frequently in both research and clinical practice. The scale is a well validated and reliable for determining change in pain over time. Pain is rated on an 11-point scale, 0-10, with 0 representing "no pain" and 10 representing "worst imaginable pain". It is well suited to this study given ease of administration in person or in online survey format. The minimum clinically important difference (MCID) for patients with knee pain secondary to osteoarthritis has been established as 2. The KOOS is also widely used in research and clinical practice, including in large-scale databases and registries. It is intended to be used in the setting of knee pain or injury that can result in post-traumatic osteoarthritis including meniscus tears. It can be used over short and long-term intervals and to asses change over time. It consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The re-test reliability has also been well established in patients with knee injuries and the MCID has been established as 8-10.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 and older
* Symptoms consistent with torn meniscus (at least one of clicking popping, giving way, pain with pivot or torque, pain that is episodic)
* Pain that can be provoked by palpitation or compression of the joint line.
* Pain located in the medial joint line that has persisted for at least 3 months.
* MRI or arthroscopic evidence of meniscal tear.
* Failed conservative treatment which has included: anti-inflammatory or other medications for pain; physical therapy; injections including corticosteroid injections and/or hyaluronic acid injections.
* This would include patients who have been told by an orthopedic surgeon that they would be a candidate for arthroscopic partial meniscectomy.

Exclusion Criteria:

* Chronically locked knee.
* Prior surgery performed on effected knee
* Assessment showing anything other than degenerative tears of the medial meniscus requiring surgical intervention.
* Recent (within 6 weeks) treatment with PRP, cortisone oral or by injection, or Hyaluronic injection.
* Any disease or condition the investigator feels would hinder treatment.
* Any contra-indication to lipoaspirate which includes: bleeding disorder, infection, pregnancy; allergy to anesthetic agents.
* Malignancy within the last 5 years.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

REFERENCES:
- [Derived] Malanga GA, Chirichella PS, Hogaboom NS, Capella T. Clinical evaluation of micro-fragmented adipose tissue as a treatment option for patients with meniscus tears with osteoarthritis: a prospective pilot study. Int Orthop. 2021 Feb;45(2):473-480. doi: 10.1007/s00264-020-04835-z. Epub 2020 Oct 7. PMID 33026537

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants were asked their age in years at the time of the intervention.
  years | 60.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Pain Scale
Description: Average knee pain between 0 (no pain) and 10 (maximum pain).
Time Frame: Baseline and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
units on a scale | -3.2 (3.6)

2. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score
Description: A scale with five subdomains that aim to capture pain, symptoms, functional limitations, and effects on quality of life caused by (in this study) meniscal injury. Each subdomain is measured from 0 (complete impairment) to 100 (no impairment). A higher score indicates less pain or better function.
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
units on a scale
  Pain | 17.5 (20.2)
  Activities of Daily Living | 17.3 (20.7)
  Symptoms | 20.5 (18.1)
  Quality of Life | 26.3 (28.9)
  Sports/Recreation | 28.4 (31.5)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03714659/Prot_SAP_000.pdf